CLINICAL TRIAL: NCT00110838
Title: Study on Omega-3 Fatty Acids and Ventricular Arrhythmia, a Parallel, Placebo-Controlled, Double Blind Intervention Study
Brief Title: SOFA: Study on Omega-3 Fatty Acids and Ventricular Arrhythmia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wageningen Centre for Food Sciences (Other)
Collaborators: SEAFOODplus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TME/C-01.07
Record Dates: First submitted 2005-05-13; First posted 2005-05-16 (Estimated); Last update posted 2006-07-21 (Estimated); Status verified 2005-05

CONDITIONS: Arrhythmia
Keywords: fish oil; n-3 fatty acids; n-3 PUFA; omega-3 fatty acids; arrhythmia; ICD; human; Patients with an implantable cardioverter defibrillator
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Dietary Supplements

INTERVENTIONS:
Procedure: Supplementation with fish oil versus placebo

SUMMARY:
The objective of the SOFA trial is to investigate whether supplemental intake of n-3 polyunsaturated fatty acids (n-3 PUFA) from fish oil can reduce the recurrence of life-threatening ventricular arrhythmias in patients with an implantable cardioverter defibrillator (ICD).

DETAILED DESCRIPTION:
Previous human observational studies and clinical trials provide strong indications that n-3 PUFA from fish can prevent cardiovascular disease. Striking is that these studies show a strong relation between n-3 PUFA and sudden death, but not between n-3 PUFA and non-fatal heart disease. Sudden death is one of the most common and often the first manifestation of coronary heart disease. The majority of sudden deaths are directly caused by acute ventricular arrhythmia. Our hypothesis is that n-3 PUFA prevents sudden death by suppressing life-threatening cardiac arrhythmia. Therefore, we investigate in a randomized controlled clinical trial whether supplemental intake of n-3 PUFA from fish can reduce the incidence of life-threatening cardiac arrhythmias. Our population consists of patients with an implantable cardioverter defibrillator (ICD), because this device records all arrhythmic events in a memory chip. As the ICD enables continuous monitoring of events in nonhospitalised patients, this population is very suitable for testing a possible antiarrhythmic effect of n-3 PUFA. The objective of the SOFA trial is to investigate the effect of fish oil on the incidence of recurrent ventricular arrhythmia in patients with an ICD. The SOFA is a randomised, parallel, placebo-controlled, double-blind intervention study which is currently being carried out in 26 cardiology centers in Europe. Five hundred forty six patients with an ICD are randomised to receive either 2g/d of fish oil or placebo oil for a period up to 12 months. The primary outcome is spontaneous ventricular tachyarrhythmias as detected by the ICD or all-cause mortality within 12 months.

ELIGIBILITY:
Inclusion Criteria:

* ICD is capable of recording ECG strips for at least 10 of its (attempted) therapeutic interventions
* 18 years or older
* written informed consent

Exclusion Criteria:

* Primary prophylactic indication
* ICD implantation as a 'bridge' to heart transplantation
* Refractory supraventricular arrhythmias with rapid ventricular rates despite antiarrhythmic therapy
* a projected lifespan of less than 1 year
* participation in another trial (during or within 30 days before SOFA)
* use of any supplemental n-3 fatty acid during the last 3 months
* intake of more than 8g of n-3 fatty acids from fish per month as judged by a fish frequency questionnaire
* pregnant women and women of childbearing potential who do not use adequate contraception
* patients known to have a history of recent drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546
Dates: Start 2001-10; Study Completion 2005-01

PRIMARY OUTCOMES:
Occurrence of appropriate ICD intervention (shock or antitachycardia pacing) for spontaneous ventricular tachyarrhythmias, or all-cause mortality

SECONDARY OUTCOMES:
All cause mortality (separately from ventricular tachyarrhythmia)
Cardiac mortality
Myocardial infarction
All arrhythmic events as documented by the ICD Core laboratory
Change in the prescription of antiarrhythmic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Evert G Schouten, MD, PhD, Study Chair — Wageningen Centre for Food Sciences
Locations (27):
- Wilhelminenspital, Vienna, Austria
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Czechia (2):
  - Interni Kardiologicka Klinika, Brno
  - Institute of Clinical and Experimental Medicine, Prague
- Germany (7):
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Klinikum Benjamin Franklin Berlin, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinikum der Friedrich-Schiller-Universitat, Jena
  - Stiftsklinik Augustinum, Munich
  - Universitatsklinikum Muenster, Münster
- Netherlands (7):
  - Academic Medical Centre Amsterdam, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - St. Antoniusziekenhuis, Nieuwegein
  - University Medical Center Rotterdam Erasmus, Rotterdam
  - University Medical Centre Utrecht, Utrecht
  - Wageningen Centre for Food Sciences, Wageningen
  - Isala Klinieken (Locatie Wezenlanden), Zwolle
- Poland (5):
  - Medical University of Gdansk, Gdansk
  - I Klinika Kardiologii, Katowice
  - Pomeranian Academy of Medicine, Szczecin
  - Instytut Kardiologii, Warsaw
  - Grochowski Hospital, Warsaw
- Centre Hospitalier Universitaire Voudois, Lausanne, Switzerland
- United Kingdom (3):
  - Queen Elizabeth Hospital, Birmingham
  - St George Hospital Medical School, London
  - Southampton General Hospital, Southampton

REFERENCES:
- [Background] Brouwer IA, Zock PL, Wever EF, Hauer RN, Camm AJ, Bocker D, Otto-Terlouw P, Katan MB, Schouten EG. Rationale and design of a randomised controlled clinical trial on supplemental intake of n-3 fatty acids and incidence of cardiac arrhythmia: SOFA. Eur J Clin Nutr. 2003 Oct;57(10):1323-30. doi: 10.1038/sj.ejcn.1601695. PMID 14506496
- [Result] Brouwer IA, Zock PL, Camm AJ, Bocker D, Hauer RN, Wever EF, Dullemeijer C, Ronden JE, Katan MB, Lubinski A, Buschler H, Schouten EG; SOFA Study Group. Effect of fish oil on ventricular tachyarrhythmia and death in patients with implantable cardioverter defibrillators: the Study on Omega-3 Fatty Acids and Ventricular Arrhythmia (SOFA) randomized trial. JAMA. 2006 Jun 14;295(22):2613-9. doi: 10.1001/jama.295.22.2613. PMID 16772624